CLINICAL TRIAL: NCT06126653
Title: A Blinded, Cross-Over Study to Evaluate the Safety and Efficacy of ARD-501 in Patients With Autism Spectrum Disorder
Brief Title: A Study to Evaluate ARD-501 in Patients With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Collaborators: Center for Psychiatry And Behavioral Medicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AARD-501.2
Record Dates: First submitted 2023-10-20; First posted 2023-11-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; High Opioid Tone; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This is a blinded, placebo controlled, cross-over trial
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Low Dose (Experimental): ARD-501 for 7 days at 0.2 mg/kg
  Interventions: Drug: Low Dose ARD-501
- Phase 2: Placebo (Placebo Comparator): Placebo for 7 days
  Interventions: Drug: Placebo
- Phase 2: High Dose (Experimental): ARD-501 for 7 days at 0.5 mg/kg
  Interventions: Drug: High Dose ARD-501
- Phase 2: Crossover Placebo to High Dose (Experimental): ARD-501 for 7 days at 0.5 mg/kg
  Interventions: Drug: High Dose ARD-501
- Phase 2: Crossover High Dose to Placebo (Placebo Comparator): Placebo for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose ARD-501 — Titratable, liquid formulation, taken orally. The intervention is given relative to the body weight of the individual. 0.2 mg/kg dosing.
  Arms: Phase 1: Low Dose
Drug: High Dose ARD-501 — Titratable, liquid formulation, taken orally. The intervention is given relative to the body weight of the individual. 0.5 mg/kg dosing.
  Arms: Phase 2: Crossover Placebo to High Dose; Phase 2: High Dose
Drug: Placebo — Titratable, liquid formulation, taken orally.
  Arms: Phase 2: Crossover High Dose to Placebo; Phase 2: Placebo

SUMMARY:
This is a blinded, placebo controlled, cross-over trial evaluating the safety of two dose-levels of ARD-501 in subjects with ASD.

DETAILED DESCRIPTION:
This study is a blinded, placebo controlled, cross-over trial evaluating the safety and efficacy of two dose levels in subjects with Autism Spectrum Disorder.

A total of up to 12 subjects will be enrolled in the clinical study.

A screening process will be initiated upon completion of the informed consent process. Subjects will be assessed for eligibility through screening tests conducted within 28 days prior to enrollment. Following completion of screening tests and confirmation of eligibility, subjects will be enrolled to complete pre-dosing requirements and questionnaires during screening window as per protocol.

There are two phases. In Phase 1, all patients will be given ARD-501 at 0.2mg/kg, dependent on their body weight (BW), for 7 days followed by a 7-day washout period. Subsequently, in Phase 2, patients will be blinded and randomized at a 1:1 ratio in two groups. Each group will be exposed to ARD-501 at 0.5mg/kg BW and placebo in alternate order. Each dosing week is followed by a 7-day washout.

All available safety and tolerability data will be evaluated throughout study conduct.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for participation in this study:

* Male and female subjects, 17-30 years of age
* Able and willing to sign consent and comply with study protocol
* Diagnostic confirmation of ASD as confirmed by gold standard clinical interview using Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) criteria and administration of the Autism Diagnostic Observation Schedule-2, Module 3 or 4.
* General good health as determined by physical exam, medical and psychiatric history and safety labs as defined by the Principal Investigator or designee.
* Male study participants who are sexually active with a female partner of childbearing potential must be surgically sterilized, or agree to use highly effective methods of birth control (defined below), and not rely on barrier methods and spermicide alone, from the time of screening until 1 week after final dose of study drug.
* Female participants of childbearing potential may be included in the study provided that they choose an effective contraception method that: 1) is not user dependent as permanent sterilization, intrauterine devices, and implants); or 2) is a user dependent short-acting hormonal method of contraception (e.g.injection, oral, transdermal, and intravaginal).

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study participation:

* Allergy or hypersensitivity to ARD-501.
* Inability to swallow study drug.
* Unstable dosing of any mood, anxiety or behavior medications in 4 weeks prior to baseline visit.
* Concomitant use of scheduled benzodiazepines, baclofen, gabapentin, pregabalin, or supplements with impact on the γ-aminobutyric acid (GABA) system.
* Concomitant use of any cannabinoid or related product.
* Any use of opioid medication
* Unstable seizure disorder as defined by any seizure in the 6 months prior to baseline visit and/or a change in any anti-convulsant drug dosing in the 60 days prior to study screen.
* Abnormal baseline safety lab assessments including, but not limited to alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than 1.5x the upper limit of normal, total bilirubin or creatinine greater than 1x the upper limit of normal, other clinically relevant lab abnormality, or abnormality in electrocardiogram (ECG), heart rate (HR), or blood pressure (BP) at screening as determined by the investigator or designee.
* History of or current abuse of drugs or alcohol including prescription medication.
* Women who are pregnant (i.e., have a positive pregnancy test), intending to become pregnant, breast feeding, or women of child-bearing potential who are unwilling to use contraception as required in the study inclusion criteria or maintain abstinence during the course of the study
* Inability to attend scheduled study visits, plans for family relocation during the study, or any other criteria that the investigator may determine to be associated with inability to complete the study
* History of major depressive disorder or history of other severe psychiatric disorders (e.g., schizophrenia or bipolar disorder) within the last 2 years.
* Suicidal ideas and behavior as assessed by the Columbia suicide severity scale (C-SSRS)
* Consumption of more than 2 units (males) or 1 unit (females) per day of alcohol during the study
* Any condition(s), including psychiatric disorders such as, but not restricted to bipolar disorders, that the investigator or primary physician believes may not be appropriate for participating the study
* Patients weighing more than 275 lb (124.7 kg)

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Assessment of the incidence of Treatment-Emergent Adverse Events (TEAE) | Baseline to Week 5
  To measure the efficacy evaluation of safety in subjects with autism spectrum disorder (ASD) by assessment of the incidence of Treatment-Emergent Adverse Events (TEAE).

SECONDARY OUTCOMES:
Assessment of change in the Clinical Global Impression - Severity/Improvement (CGI-S/I) scale | Baseline to Week 5
  To evaluate efficacy in subjects with ASD on the Clinical Global Impression - Severity/Improvement (CGI-S/I) scale
Assessment of change on the Social Responsiveness Scale, Second Edition (SRS™-2, version-adjusted for age) | Baseline to Week 5
  To evaluate efficacy in social responsiveness in subjects with ASD on the Social Responsiveness Scale, Second Edition (SRS™-2, version-adjusted for age).

OTHER OUTCOMES:
Assessment of change in Gastrointestinal Severity Index (GSI) | Baseline to Week 5
  To evaluate the efficacy of improvement in the gastrointestinal severity as assessed by the Gastrointestinal Severity Index (GSI)
Assessment of change in Pain Detection Threshold (PDT) and Pain Tolerating Threshold (PTT) as measured during the Cold Pressor Test | Baseline to Week 5
  To evaluate efficacy of improvement or change in Pain Detection Threshold (PDT) and Pain Tolerating Threshold (PTT) as measured during the Cold Pressor Test
Assessment of change on the Adaptive Behavior Assessment System (ABAS-3) | Baseline to Week 5
  To evaluate efficacy in adaptive behavior as assessed by change in the Adaptive Behavior Assessment System (ABAS-3)
Assessment of change on the Aberrant Behavior Checklist, Second Edition (ABC-2) | Baseline to Week 5
  To evaluate efficacy in deviant interactions as assessed by change in the Aberrant Behavior Checklist (ABC-2)
Assessment of change on the Difficulties in Emotion Regulation Scale (DERS) | Baseline to Week 5
  To evaluate efficacy in emotional response and management as assessed by change in the Difficulties in Emotion Regulation Scale (DERS)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Psychiatry and Behavioral Medicine Inc, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No